CLINICAL TRIAL: NCT06225791
Title: Implementation Research to Accelerate Multiple Micronutrient Supplementation During Pregnancy in Indonesia
Brief Title: Antenatal Multiple Micronutrient Supplementation (MMS) in Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Indonesia University (Other); Hasanuddin University (Other); Universitas Airlangga (Other); Vitamin Angels (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00016428 / MOD00004017
Record Dates: First submitted 2023-12-19; First posted 2024-01-26 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Nutrient Deficiency
Keywords: multiple micronutrient supplementation (MMS); pregnancy; behavior change; packaging; antenatal care (ANC)

STUDY DESIGN:
Intervention Model Description: MMS will be implemented across 13 districts in Indonesia. In each of the 8 high-intensity evaluation districts and 5 moderate-intensity evaluation districts, 3 study arms/sub-districts have been purposively selected (total n = 24 sub-districts).
  * Arm/sub-district 1: Provision of 90-count bottles x 2, with standard MMS delivery strategies and MMS orientation
  * Arm/sub-district 2: Provision of 90-count bottles x 2, with enhanced MMS deliveries strategy (3 with MMS orientation with BCC; 5 with MMS orientation with expanded BCC)
  * Arm/sub-district 3: Provision of 180-count bottles x 1, with enhanced MMS delivery strategy (3 with MMS orientation with BCC; 5 with MMS orientation with expanded BCC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard MMS delivery with two 90-count bottles (No Intervention): Pregnant women are provided with two 90-count bottles of MMS at two different time points during pregnancy, along with standard MMS delivery strategy (MMS orientation only). (1 sub-district within each of the 13 districts with high- or moderate-intensity evaluation).
- Enhanced MMS delivery with two 90-count bottles (Active Comparator): Pregnant women are provided with two 90-count bottles of MMS at two different time points during pregnancy, along with enhanced MMS delivery strategy (5 districts with MMS orientation with BCC; 8 districts with MMS orientation with expanded BCC). (1 sub-district within each of the 13 districts with high- or moderate-intensity evaluation).
  Interventions: Behavioral: MMS (90x2) + BCC or expanded BCC
- Enhanced MMS delivery with one 180-count bottle (Active Comparator): Pregnant women are provided with one 180-count bottle of MMS along with enhanced MMS delivery strategy (5 districts with MMS orientation with BCC; 8 with MMS orientation with expanded BCC). (1 sub-district with each of the 13 districts with high- or moderate-intensity evaluation).
  Interventions: Behavioral: MMS (180x1) + BCC or expanded BCC

INTERVENTIONS:
Behavioral: MMS (90x2) + BCC or expanded BCC — Provision of 90-count bottles x 2, with enhanced MMS delivery strategy (5 districts with MMS orientation with BCC; 8 districts with MMS orientation with expanded BCC)
  Arms: Enhanced MMS delivery with two 90-count bottles
Behavioral: MMS (180x1) + BCC or expanded BCC — Provision of 180-count bottles x 1, with enhanced MMS delivery strategy (5 districts with MMS orientation with BCC; 8 districts with MMS orientation with expanded BCC)
  Arms: Enhanced MMS delivery with one 180-count bottle

SUMMARY:
The objective of this research is to understand how antenatal multiple micronutrient supplements (MMS) can be effectively implemented and scaled within the Indonesian national health system context to support improved maternal nutrition and birth outcomes. Formative research has been conducted to design the implementation strategies that will be tested in this second phase of the study. The objectives are to:

* Examine different MMS delivery strategies (i.e., packaging strategies and behavior change communication (BCC) strategies) in relation to MMS adherence.
* Assess acceptability, feasibility, fidelity, and coverage of MMS program implementation within antenatal care services (ANC)

DETAILED DESCRIPTION:
The study will utilize qualitative and quantitative methods to:

* Test different MMS delivery strategies (bottle count [90 vs. 180 tablets] and communication strategies [BCC vs. expanded BCC vs. MMS orientation only]) for enhancing supplementation consumption - measured as coverage and adherence.
* Assess acceptability, feasibility, and fidelity of MMS program implementation within antenatal care services (ANC)

More specifically, the investigators will implement and evaluate different MMS packaging (90 count bottle vs 180-count bottle) strategies and behavior change communication (BCC) strategies. The 3 BCC approaches are further described below.

* BCC, BCC without Interpersonal Communication (IPC) strategy is a briefer more basic approach that hopes to improve health care providers knowledge about MMS and the providers ability to communicate with pregnant women. This approach will be rolled out by training one district-level facilitator in each district to become a trainer who will be responsible for training health providers in the corresponding study sub-districts.
* Expanded BCC ('BCC with Interpersonal Communication [IPC]') needs more intensive training of master trainers to train health care providers and focuses more on the counselling skills portion. The BCC without IPC is more feasible to implement within the existing system, the investigators anticipate that the BCC with IPC achieve better behavior change results.
* MMS Orientation: Women in the control group will receive the existing standard of counselling care. The providers will not be given any sort of training on counselling. Due to the fact that MMS is a new product that the providers will be providing pregnant women, all health care providers will receive a standard MMS orientation so providers are comfortable with the new supplement.

The study will be conducted in 25 districts representing the western, central, and eastern regions of Indonesia, Indonesia's socio-cultural diversity, and varying capacity of ANC systems across districts. After selection, the 25 districts were divided to receive high-intensity (8 districts), moderate-intensity (5 districts), or low-intensity (12 districts) evaluation activities with those exposed to high-intensity evaluation efforts having comprehensive individual-level data collected by study employed data collectors while the low-and moderate-intensity district data collection efforts are being done within the context of the existing health system.

1. High intensity evaluation areas (8 districts) Evaluation of MMS acceptability, coverage, adherence, feasibility, and fidelity will include data collection from health professionals and pregnant women by study data collectors, and by ANC monitoring activities.
2. Moderate intensity evaluation areas (5 districts) Evaluation of ANC records with aggregate coverage and adherence numbers will be shared with investigators. In addition, data collectors will collect MMS acceptability, feasibility, and fidelity data within 2 of those 5 districts.
3. Low intensity evaluation area (12 districts) Evaluation of ANC records with aggregate coverage and adherence numbers will be shared with investigators. In addition, a household coverage survey will be administered in a subset of districts (n=6) post-intervention to examine MMS acceptability, adherence, coverage, and implementation feasibility and fidelity. The coverage survey will be designed after 6 months of implementation and will be submitted as a separate application to the Johns Hopkins Bloomberg School of Public Health Institutional Review Board, and a separate entry into Clinicaltrials.gov.

Within the 8 high-intensity districts and 5 moderate-intensity districts that are the subject of this Clinicaltrials.gov submission, the study will utilize a three-arm cluster randomized design (with sub-district health center as the unit of randomization).

ELIGIBILITY:
Inclusion Criteria for 3,360 pregnant women (PW) enrolled from 8 high-intensity evaluation districts (sample group 1)

* Enrolled in ANC 1 through government health facilities.
* Received MMS at ANC 1
* Gestational age at ANC 1 ≤ 20 weeks (verified by health professionals)
* Consent provided to participate in the study.

Exclusion Criteria for 3,360 pregnant women (PW) enrolled from 8 high-intensity evaluation districts (sample group 1)

* PW with complicated pregnancy complications (e.g., thalassemia, hemochromatosis,)
* PW planning to move outside study district during study period.

Inclusion Criteria for 72 PW / recently delivered women participating in in-depth interviews (IDI) only (sample group 2)

* Enrolled in ANC 1 through government health facilities.
* Received MMS at ANC 1
* Gestational age at ANC 1 ≤ 20 weeks (verified by health professionals)
* Consent provided to participate in qualitative component of study.
* Received MMS for at least 3 months.
* Attended > 2 ANC visits.
* < 4 weeks post-partum

Exclusion Criteria for 72 PW / recently delivered women participating in in-depth interviews (IDI) only (sample group 2)

* Enrolled in Sample 1
* Women who are more than 4 weeks postpartum.

Inclusion Criteria for 180 healthcare providers participating in focus group discussions (FGDs) (sample group 3)

* Government health workers who provide ANC services (e.g., midwives, general practitioners, and nutritionists)
* Government health facility management staff (e.g., Head of Puskesmas Community Health Clinic, Coordinating Midwife, Head of Pharmacy)
* Willing to give consent to participate in the FGD.

Exclusion Criteria for 180 healthcare providers participating in FGDs (sample group 3) • Healthcare Providers who have already participated in a FGD will not be eligible to participate in another FGD

Inclusion Criteria for 76 government decision-makers participating in FGD or IDI (sample group 4)

* District-, provincial-, or national-level decision-makers working in nutrition, maternal, newborn and child health, or pharmaceutical roles associated with the antenatal care system in Indonesia.
* Willing to give consent to participate in the FGD or IDI.

Exclusion Criteria for 76 government decision-makers participating in FGD or IDI (sample group 4)

• None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5384 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
MMS Adherence (amount) | Post-enrollment up to 3 months, Post-pregnancy up to 4 weeks
  The number of MMS tablets (from a total possible 180 tablets) a pregnant woman consumes (sample group 1).
MMS Adherence (frequency) | Post-enrollment up to 3 months, Post-pregnancy up to 4 weeks
  The frequency of which MMS tablets are consumed by a pregnant woman. (sample group 1)

SECONDARY OUTCOMES:
MMS Acceptability among Pregnant Women | Post-enrollment up to 3 months, Post-pregnancy up to 4 weeks
  The proportion of pregnant women (sample group 1 and 2) who agree with domain-specific statements which reflect different aspects of MMS acceptability (MMS packaging, MMS physical properties, MMS side effects, and MMS counseling using The Theoretical Framework of Acceptability uses a 5-point Likert scale where 5 is "strongly agree" and 1 is "strongly disagree". Score range 5-35, a higher score reflects higher acceptability.
MMS Acceptability among Health Providers assessed by focus group discussions | 6 months, 12 months
  Healthcare provider acceptability of MMS across multiple domains (e.g., feasibility of delivering counseling and packaging, time burden) (sample group 3). Measured via focus group discussions at two time points during the study (middle and end).
Fidelity of providing MMS among Health Providers as assessed by focus group discussions | 6 months, 12 months
  Administration of an observation checklist (sample group 3),measured via focus group discussions at two time points during the study (middle and end)

OTHER OUTCOMES:
Number of pregnant women being given 180 tablets of MMS | Monthly up to 18 months
  MMS coverage as assessed by the number of pregnant women being given 180 tablets of MMS as compared to the estimated number of pregnant women in the population (e.g., within the 24 study sub-districts) via routine data collection from facility to district health office (aggregate data).
Number of MMS tablets consumed | Monthly up to 18 months
  MMS adherence as assessed by the number of MMS tablets (from a total of 180 tablets) women who receive MMS are consuming. Routine Data Collection (aggregate data) from facility to district health office.

CONTACTS AND LOCATIONS:
Overall Officials: Endang Achadi, PhD, Principal Investigator — Indonesia University; Kristin Hurley, PhD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Universitas Indonesia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No